CLINICAL TRIAL: NCT00997503
Title: TAXUS Libertē Post Approval Study: A U.S. Post-Approval Study of the TAXUS® Liberté® Paclitaxel-Eluting Coronary Stent System
Brief Title: TAXUS Libertē Post Approval Study
Status: Completed | Type: Observational
Sponsor: Boston Scientific Corporation (Industry)
Collaborators: Eli Lilly and Company (Industry); Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Other Study IDs: H7T-MC-TADN; S2035 (Other: Boston Scientific)
Record Dates: First submitted 2009-10-15; First posted 2009-10-19 (Estimated); Results first posted 2015-04-13 (Estimated); Last update posted 2015-08-07 (Estimated); Status verified 2015-03

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Prasugrel Hydrochloride; Aspirin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: TAXUS Liberté Paclitaxel-Eluting Coronary Stent — The TAXUS Liberté Paclitaxel-Eluting Coronary Stent System is a device/drug combination product comprised of two regulated components: a device (Liberté Coronary Stent System) and a drug product (a formulation of paclitaxel contained in a polymer coating).The polymer coating serves as a carrier system to provide uniform and controlled biphasic release of the drug into the vessel wall once the stent is deployed.
Drug: prasugrel — 10mg or 5mg, oral, once daily as maintenance dose through 30-months following index procedure
  Other Names: Effient
Drug: placebo — Oral placebo to match both 10mg and 5mg prasugrel tablets.
Drug: aspirin — Oral, as prescribed by physician through end of study.
  .

SUMMARY:
The TAXUS Libertē Post-Approval Study is an FDA-mandated prospective, multi-center study designed to collect real-world safety and clinical outcomes in approximately 4,200 patients receiving one or more TAXUS Liberté Paclitaxel-Eluting Stents and prasugrel as part of a dual antiplatelet therapy (DAPT) drug regimen.

This study will also contribute patient data to an FDA-requested and industry-sponsored research study that will evaluate the optimal duration of dual antiplatelet therapy (DAPT Study).

DETAILED DESCRIPTION:
The TAXUS Libertē Post-Approval Study is an FDA-mandated prospective, multi-center study designed to collect real-world safety and clinical outcomes in approximately 4,200 patients receiving one or more TAXUS Liberté Paclitaxel-Eluting Stents and prasugrel as part of a dual antiplatelet therapy (DAPT) drug regimen. This is a consecutively-enrolled study with patient follow-up through 3 years post index procedure. This study also will contribute patient data to an FDA-requested and industry-sponsored research study that will evaluate the optimal duration of dual antiplatelet therapy (DAPT Study). To facilitate this patient data contribution, patients will be assigned to patient groups based upon their co-morbidities and stented lesions identified post index procedure.

All enrolled patients who have been treated with the TAXUS Liberté Stent will be assigned to 12 months of open-label prasugrel treatment and aspirin. Upon completion of the open-label period, patients who are clear of events at 12 months post index procedure will be randomized 1:1 to either a placebo or prasugrel for an additional 18 months of treatment. All patients will receive aspirin therapy throughout the course of the study.

ELIGIBILITY:
Enrollment Inclusion Criteria

* Patient is > 18 years of age.
* Consecutive patients who have signed an Informed Consent Form, who do not otherwise meet applicable exclusion criteria, and who are eligible to receive a TAXUS Liberté Stent and the study required DAPT will be evaluated for enrollment in this study.

Enrollment Exclusion Criteria

* Patient with known hypersensitivity to paclitaxel or structurally related compounds.
* Patient with known hypersensitivity to the polymer or any of its individual components.
* Patient judged to have a lesion that prevents complete inflation of an angioplasty balloon or proper placement of the stent or delivery device.
* Patient who cannot receive the protocol required dual antiplatelet therapy.
* Patient on warfarin or similar anticoagulant therapy.
* Patient with known pregnancy.
* Planned surgery necessitating discontinuation of antiplatelet therapy(> 14 days)within the 30-months following enrollment.
* Current medical condition with a life expectancy of less than 3 years.
* Patient currently enrolled in another device or drug study whose protocol specifically excludes concurrent enrollment or that involves blinded placement of a drug-eluting stent other than the TAXUS Liberté Stent.
* Patient judged unable to cooperate with prolonged DAPT.
* Patient unable to give informed consent.
* Patient judged inappropriate for randomization due to other condition requiring chronic thienopyridine use.
* Patient treated with both a drug-eluting stent and a bare-metal stent during the index procedure.
* Patient who experienced a prior transient ischemic attack (TIA) or a prior stroke.
* Patient requiring chronic daily use (greater than 2 consecutive weeks) of non-steroidal anti-inflammatory drugs (NSAIDs) with the exception of aspirin. Occasional use of NSAIDs on an as needed or "prn" schedule is not exclusionary.
* Patient with active pathological bleeding (such as peptic ulcer or intracranial hemorrhage).

Additional Exclusion Criteria (applicable only after patient enrollment has reached approximately 3600)

* Patient who experienced a myocardial infarction (MI) within 72 hours prior to the index procedure.
* Patient with a history of (includes current) left main coronary artery disease.
* Patient who requires stenting of > 1 vessel with a TAXUS Liberté stent during the index procedure.
* Patient who requires stenting of > 2 vessels during the index procedure.
* Patient who requires a staged procedure within 6-weeks following the index procedure, in whom > 1 vessel was stented during the index procedure.
* Patient with cardiogenic shock.
* Patient with acute or chronic renal dysfunction (serum creatinine >3.0 mg/dl or patient receiving dialysis).
* Target Lesion that meets any of the following criteria:

  * Located within a saphenous vein graft or an arterial graft
  * Chronic total occlusion
  * Restenosis from a previously implanted drug-eluting or bare-metal stent
  * Previous use of intravascular brachytherapy in target vessel
  * Lesion involves a bifurcation
  * Lesion is ostial in location
  * Severe tortuosity in the target lesion or target vessel proximal to the target lesion
  * Moderate or severe calcification by visual estimate in the target lesion or target vessel proximal to the target lesion
  * RVD < 2.5 mm or RVD > 3.75 mm
  * Lesion length > 28 mm

Randomization Inclusion Criteria (12-months):

* Patient is "12-Month Clear," which is defined as patients enrolled in the study who are free from all death, MI, stroke, repeat coronary revascularization, stent thrombosis and major bleeding (severe or moderate by GUSTO classification) 12 months after stent implantation and who are compliant with 12 months of DAPT following stent implantation. Exceptions to this rule are: Patients who experience repeat PCI, stent thrombosis and/or myocardial infarction occurring within 6 weeks after the index procedure will not be excluded from the definition of 12-Month Clear.
* Patient was compliant with DAPT during the first 12 months of the study. Compliance is defined as the patient taking between 80% and 120% of prasugrel in the 0-6 month and 6-12 month periods without an interruption of therapy longer than 14 days. Compliance at both time points is required to be considered 12-Month Clear.

Randomization Exclusion Criteria (12-months):

* Known pregnancy.
* Patient switched from prasugrel to other thienopyridine after discharge from index hospitalization.
* Patient switched maintenance dose of prasugrel (such as 10mg to 5mg; or 5mg to 10mg) within 6-months prior to randomization.
* Percutaneous coronary intervention or cardiac surgery between 6 weeks post index procedure and randomization.
* Planned surgery necessitating discontinuation of antiplatelet therapy (> 14 days) within the 21 months following randomization.
* Patients on warfarin or similar anticoagulant therapy.
* Current medical condition with life expectancy of less than 3 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All-comers study with follow-up through 3 years.
Sampling Method: Non-Probability Sample
Enrollment: 4199 (Actual)
Dates: Start 2009-12; Primary Completion 2013-03 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David P Lee, MD, Principal Investigator — Stanford University; Kirk N Garratt, MD, Principal Investigator — Lenox Hill Hospital; Peter M Maurer, MPH, Study Director — Boston Scientific Corporation
Locations (82):
- United States (82):
  - Advanced Cardiac Specialists, Mesa, Arizona
  - NEA Baptist Memorial Hospital, Jonesboro, Arkansas
  - St. Bernard's Medical Center, Jonesboro, Arkansas
  - Baptist Health Medical Center, Little Rock, Arkansas
  - Bakersfield Memorial Hospital, Bakersfield, California
  - Bakersfield Heart, Bakersfield, California
  - Mercy General Hospital, Sacramento, California
  - Alvarado Hospital, San Diego, California
  - Stanford University Medical Center, Stanford, California
  - Torrance Memorial Medical Center, Torrance, California
  - St. Anthony Central Hospital, Denver, Colorado
  - Medical Center of the Rockies (Loveland), Loveland, Colorado
  - St. Vincent's Medical Center, Bridgeport, Connecticut
  - Christiana Hospital, Newark, Delaware
  - JFK Medical Center, Atlantis, Florida
  - North Florida Regional Medical Center, Gainesville, Florida
  - Baptist Medical Center, Jacksonville, Florida
  - Memorial Hospital Jacksonville/ Orange Park Medical Center, Jacksonville, Florida
  - Holmes Regional Medical Center, Melbourne, Florida
  - Florida Hospital, Orlando, Florida
  - Baptist Hospital, Pensacola, Florida
  - Sacred Heart Hospital, Pensacola, Florida
  - Bayfront Medical Center, St. Petersburg, Florida
  - Martin Memorial Medical Center, Stuart, Florida
  - University Community Hospital, Tampa, Florida
  - Kaiser Foundation Hospitals, Honolulu, Hawaii
  - Kootenai Medical Center, Coeur d'Alene, Idaho
  - MacNeal Hospital, Berwyn, Illinois
  - Jesse Brown VA Medical Center, Chicago, Illinois
  - IU Health North Medical Center, Carmel, Indiana
  - Indiana Heart Hospital, Indianapolis, Indiana
  - King's Daughters Medical Center- Kentucky Heart Institute, Ashland, Kentucky
  - St. Joseph Hospital, Lexington, Kentucky
  - Christus St. Frances Cabrini Hospital, Alexandria, Louisiana
  - Cardiovascular Research, LLC, Shreveport, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Central Maine Medical Center, Lewiston, Maine
  - Genesys Regional Medical Center, Grand Blanc, Michigan
  - Ingham Regional Medical Center, Lansing, Michigan
  - Mid Michigan Medical Center, Midland, Michigan
  - St. Mary's Medical Center, Mount Pleasant, Michigan
  - Northern Michigan Hospital, Petoskey, Michigan
  - Covenant Medical Center, Saginaw, Michigan
  - Lakeland Hospital at St. Joseph, Saint Joseph, Michigan
  - Providence Hospital, Southfield, Michigan
  - North Memorial Medical Center, Minneapolis, Minnesota
  - United Heart and Vascular Clinic, Saint Paul, Minnesota
  - Memorial Hospital at Gulfport, Gulfport, Mississippi
  - North Mississippi Medical Center, Tupelo, Mississippi
  - Freeman West Hospital, Joplin, Missouri
  - Cox Medical Centers, Springfield, Missouri
  - St. John's Mercy Medical Center, St Louis, Missouri
  - Our Lady of Lourdes Medical Center, Camden, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Jersey Shore University Medical Center, Neptune City, New Jersey
  - Heart Hospital of New Mexico, Albuquerque, New Mexico
  - Maimonides Medical Center, Brooklyn, New York
  - Lenox Hill Hospital, New York, New York
  - Columbia University/ New York Presbyterian Hospital, New York, New York
  - St. Elizabeth Medical Center, Utica, New York
  - Gaston Memorial Hospital, Gastonia, North Carolina
  - Wake Medical Center, Raleigh, North Carolina
  - Ohio State University Medical Center, Columbus, Ohio
  - Med Central Health System- Mid Ohio Heart Clinic, Mansfield, Ohio
  - St. Vincent Mercy Medical Center, Toledo, Ohio
  - University of Oklahoma Health Science Center, Oklahoma City, Oklahoma
  - Oklahoma Heart Hospital, Oklahoma City, Oklahoma
  - Conemaugh Valley Memorial Hospital, Johnstown, Pennsylvania
  - Presbyterian University of Pennsylvania Medical Center, Philadelphia, Pennsylvania
  - Palmetto Richland Memorial Hospital, Columbia, South Carolina
  - Sisters of Charity Providence Hospital, Columbia, South Carolina
  - Grand Strand Regional Medical Center, Myrtle Beach, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Avera Heart Hospital of South Dakota, Sioux Falls, South Dakota
  - Jackson Madison County General Hospital, Jackson, Tennessee
  - Baylor Jack and Jane Hamilton Heart and Vascular Hospital, Dallas, Texas
  - Doctors Hospital at Renaissance/ McAllen Heart Hospital, Edinburg, Texas
  - Michael E. DeBakey VA Medical Center, Houston, Texas
  - Kingwood Medical Center, Kingwood, Texas
  - Methodist Texsan Hospital, San Antonio, Texas
  - Cardiovascular Associates of East Texas Medical Center, Tyler, Texas
  - Meriter Hospital, Inc., Madison, Wisconsin

REFERENCES:
- [Background] Ellis SG, Vandormael MG, Cowley MJ, DiSciascio G, Deligonul U, Topol EJ, Bulle TM. Coronary morphologic and clinical determinants of procedural outcome with angioplasty for multivessel coronary disease. Implications for patient selection. Multivessel Angioplasty Prognosis Study Group. Circulation. 1990 Oct;82(4):1193-202. doi: 10.1161/01.cir.82.4.1193. PMID 2401060
- [Result] Lee DP, Paulus R, Giri K, Carr J, Baran KW, Hassel D, Winters KJ, Christen T, Dawkins KD, Garratt KN. TCT-167 Primary endpoint results of the TAXUS Libertē post-approval study. Journal of the American College of Cardiology. 2013;62:B54-B54
- [Result] Garratt, KN, Lambert C, Kabour A, Stewart M, Hall P, Phillips WJ, Winters KJ, Christen T, Dawkins KD, Lee DP TCT-148 TAXUS Liberté PES With ASA + Prasugrel Is Associated With Low TVF, Bleeding And Adverse Event Rates Among Diabetic Patients With "On-Label" Stent Indications. Journal of the American College of Cardiology, 2013; 62 (18_S1): B47-B47.
- [Derived] Garratt KN, Weaver WD, Jenkins RG, Pow TK, Mauri L, Kereiakes DJ, Winters KJ, Christen T, Allocco DJ, Lee DP. Prasugrel plus aspirin beyond 12 months is associated with improved outcomes after TAXUS Liberte paclitaxel-eluting coronary stent placement. Circulation. 2015 Jan 6;131(1):62-73. doi: 10.1161/CIRCULATIONAHA.114.013570. Epub 2014 Nov 16. PMID 25400062

RESULTS

PARTICIPANT FLOW:
Groups:
- TAXUS Libertē: Overall Enrolled Population: Overall enrolled population of patients: received at least one TAXUS Liberté Paclitaxel-Eluting Coronary Stent System in routine clinical practice, in conjunction with the use of prasugrel and aspirin.
Period: Overall Study
Arm/Group | TAXUS Libertē: Overall Enrolled Population
Started | 4199
12 Months | 4059 (4059 subjects evaluable at 12-months (cardiac death/MI within 365 days or completed follow-up))
Completed | 3926
Not Completed | 273
Not completed — Death | 53
Not completed — Withdrawal by Subject | 76
Not completed — Lost to Follow-up | 33
Not completed — Adverse Event | 3
Not completed — Physician Decision | 10
Not completed — Missed 12-month follow-up | 85
Not completed — Other reason | 13

BASELINE CHARACTERISTICS:
Groups:
- TAXUS Liberté Post-Approval Study Enrolled Population: Overall enrolled population of patients: received at least one TAXUS Liberté Paclitaxel-Eluting Coronary Stent System in routine clinical practice, in conjunction with the use of prasugrel and aspirin.
Arm/Group | TAXUS Liberté Post-Approval Study Enrolled Population
Number analyzed (Participants) | 4199
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.8 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1161
  Male | 3038
Race/Ethnicity, Customized [Number; unit: participants] — Some participants may be allocated to greater than one category.
  participants
    Hispanic or Latino | 181
    Caucasian | 3623
    Asian | 23
    Black, or African Heritage | 323
    Native Hawaiian or Other Pacific Islander | 8
    American Indian or Alaska Native | 16
    Other | 43
Region of Enrollment [Number; unit: participants]
  United States | 4199
Weight [Mean (Standard Deviation); unit: kilograms] | 92.9 (20.7)
Smoking Status [Number; unit: participants]
  Current | 1272
  Previous | 1451
  Never | 1387
  Unknown | 89
History of Hyperlipidemia Requiring Medication [Number; unit: participants] | 2950
History of Hypertension Requiring Medication [Number; unit: participants] | 3130
Diabetic (Medically Treated) [Number; unit: participants] | 1289
Family History of Coronary Artery Disease (CAD) [Number; unit: participants] | 2466
History of Atrial Fibrillation [Number; unit: participants] | 143
History of Coronary Artery Bypass Graft (CABG) [Number; unit: participants] | 559
History of Percutaneous Coronary Intervention (PCI) [Number; unit: participants] | 1411
History of Congestive Heart Failure (CHF) [Number; unit: participants] | 254
Current Stable Angina [Number; unit: participants] — Canadian Cardiology Society Classification (CCSC)
  participants | 1320
Current Unstable Angina [Number; unit: participants] | 1385
Current Silent Ischemia [Number; unit: participants] | 310
Current Myocardial Infarction (MI) [Number; unit: participants] | 1040
Experiencing Cardiogenic Shock [Number; unit: participants] — A clinical state of hypoperfusion characterized by systolic pressure <80 mm Hg and/or central filling pressure >20 mm Hg, or cardiac index <1.8 liters/minute/m2 where there is evidence of insufficient end organ profusion. Shock is also considered present if intravenous inotropes and/or intra-aortic balloon pump are needed to maintain a systolic blood pressure >80 mm Hg and a cardiac index >1.8 liters/minute/ m2.
  participants | 17
History of Multivessel Disease [Number; unit: participants] — The presence of a greater than 50% diameter stenosis in 2 or 3 major epicardial coronary vessels or bypassed branches.
  participants | 1464
History of Left Main Disease [Number; unit: participants] | 155
History of Transient Ischemic Attack (TIA) [Number; unit: participants] | 4
History of Stroke [Number; unit: participants] | 4
Current Renal Dysfunction [Number; unit: participants] | 185
History of Peripheral Vascular Disease [Number; unit: participants] | 284
History of Major Bleeding [Number; unit: participants] | 32
De Novo Lesion [Number; unit: lesions] — A coronary lesion not previously treated.
  lesions | 5421
Culprit Lesion for ST Elevation Myocardial Infarction (STEMI) [Number; unit: lesions] | 386
Restenosis [Number; unit: lesions]
  Restenosis - Drug Eluting Stent (DES) | 168
  Restenosis - Bare Metal Stent (BMS) | 82
  Restenotic Lesion (No Stent) | 31
Chronic Total Occlusion [Number; unit: lesions] — Lesion that has been totally occluded for three or more months and with a documented TIMI flow of 0.
  lesions | 70
Ostial Lesion [Number; unit: lesions] — Lesions involving the origin of the coronary artery within the first 3 mm.
  lesions | 216
Post Brachytherapy [Number; unit: lesions] | 5
Bifurcated Lesion [Number; unit: lesions] — Lesion where a branch vessel of medium or large size originates.
  lesions | 336
Reference Vessel Diameter (RVD) [Mean (Standard Deviation); unit: millimeters] | 2.99 (0.5)
Lesion Length [Mean (Standard Deviation); unit: millimeters] — Measured as distance from the proximal to the distal shoulder in the view that demonstrates the stenosis in its most elongated projection; lesion length is recorded as discrete (<10 mm), tubular (10-20 mm), and diffuse (>20 mm).
  millimeters | 16 (9.5)
Pre-Procedure Thrombolysis In Myocardial Infarction (TIMI) Flow [Number; unit: lesions] — TIMI 0 No perfusion.
  TIMI 1 Penetration with minimal perfusion. Contrast fails to opacify the entire bed distal to the stenosis of the duration of the cine run.
  TIMI 2 Partial perfusion. Contrast opacifies the entire coronary bed distal to the stenosis. However, the rate of entry and/or clearance is slower in the coronary bed distal to the obstruction than in comparable areas not perfused by the dilated vessel.
  TIMI 3 Complete perfusion. Filling and clearance of contrast equally rapid in the coronary bed distal to stenosis as in other coronary beds.
  lesions
    0 | 501
    1 | 197
    2 | 679
    3 | 4283
Lesion Classification: American College of Cardiology (ACC)/ American Heart Association (AHA) [Number; unit: lesions] — Please note the reference section for further definition of the lesion classification.
  lesions
    Type A | 1132
    Type B1 | 2298
    Type B2 | 1162
    Type C | 1068
Lesion Calcification [Number; unit: lesions] — Readily apparent densities seen within the artery wall and site of lesion either as an X-ray absorbing mass or as an echogenic and shadow generating mass in IVUS imaging; these can be classified as little/none, moderate, or severe.
  lesions
    None | 3630
    Mild | 1398
    Moderate | 482
    Severe | 150
Pre-Procedure Target Lesion Percent Diameter Stenosis (%DS) [Mean (Standard Deviation); unit: percemt] | 85.3 (11.7)
Vessel Tortuosity [Number; unit: lesions]
  None | 3912
  Mild | 1261
  Moderate | 431
  Severe | 56
Lesion Location (Vessel) [Number; unit: lesions]
  Right Coronary Artery (RCA) | 1943
  Left Anterior Descending (LAD) Coronary Artery | 2198
  Left Circumflex (LCX) Coronary Artery | 1306
  Left Main (LM) Coronary Artery | 46
  Arterial or Vein Graft | 167
Thrombus Present (Pre-Procedure) [Number; unit: lesions]
  Yes | 478
  Possibly | 273
  No | 4840
  Unknown | 69
Acute Coronary Syndrome (ACS) Present [Number; unit: procedures] — * Subjects may have more than 1 procedure (enrollment and staged)
  * ACS is defined as ischemic symptoms occurring at rest and lasting 10 minutes or more and occurring within 72 hours before index procedure and either ST-segment deviation of 1 mm or more or elevated levels of a cardiac biomarker of necrosis (CK-MB or troponin T or I greater than the upper limit of normal. If CK-MB or troponin is not available, total CK >2 times upper limit of normal). Subjects with STEMI can be enrolled at any time, and will be classified as ACS and therefore complex, within 14 days after onset of symptoms.
  procedures | 1194
Pre-dilatation Performed [Number; unit: procedures] | 3044
Number of Lesions Treated Per Patient [Mean (Standard Deviation); unit: lesions] | 1.3 (0.7)
Number of Vessels Treated Per Patient [Mean (Standard Deviation); unit: vessels] | 1.1 (0.4)
Study Stents Implanted Per Patient [Mean (Standard Deviation); unit: stents] | 1.5 (0.8)
Post-Procedure Thrombolysis In Myocardial Infarction (TIMI) Flow [Number; unit: lesions] — TIMI 0 No perfusion.
  TIMI 1 Penetration with minimal perfusion. Contrast fails to opacify the entire bed distal to the stenosis of the duration of the cine run.
  TIMI 2 Partial perfusion. Contrast opacifies the entire coronary bed distal to the stenosis. However, the rate of entry and/or clearance is slower in the coronary bed distal to the obstruction than in comparable areas not perfused by the dilated vessel.
  TIMI 3 Complete perfusion. Filling and clearance of contrast equally rapid in the coronary bed distal to stenosis as in other coronary beds.
  lesions
    0 | 0
    1 | 1
    2 | 42
    3 | 5617
Post-Procedure Target Lesion Percent Diameter Stenosis (%DS) [Mean (Standard Deviation); unit: percentage of diameter stenosis] | 1.3 (4.2)
Thrombus Present (Post-Procedure) [Number; unit: lesions]
  Yes | 27
  Possibly | 45
  No | 5588

OUTCOME MEASURES:

1. Primary Outcome: Cardiac Death or Myocardial Infarction
Description: Cardiac death or myocardial infarction in the TAXUS Liberte Post-Approval Study enrolled population. For pooled data from the TAXUS Liberté and TAXUS Express patient populations, please see the citations.
Time Frame: 12 months
Population: There were 140 patients that were not eligible for the 12-month analyses, as they did not meet the following criteria: either a minimum number of days of follow-up of 335 days or an endpoint event up to 365 days post-stent implant procedure.
Measure: Number; unit: percentage of participants
Groups:
- TAXUS Libertē Post-Approval Study Enrolled Population: There were a total of 4,199 patients in the TAXUS Libertē Post-Approval Study that received at least one TAXUS Liberte stent.
Arm/Group | TAXUS Libertē Post-Approval Study Enrolled Population
Number analyzed (Participants) | 4059
percentage of participants | 2.1

2. Secondary Outcome: Incremental Rate of Stent Thrombosis (Protocol Definition)
Description: Stent Thrombosis (protocol definition):
  The occurrence of any of the following:
  1. Clinical presentation of acute coronary syndrome with angiographic evidence of stent thrombosis:
     Angiographic documentation of acute complete occlusion (TIMI flow 0 or 1) of a previously successfully treated artery (TIMI flow 2 to 3 immediately after stent placement and diameter stenosis less than or equal to 30%) and/or Angiographic documentation of a flow limiting thrombus within or adjacent to a previously successfully treated lesion
  2. Acute MI in the distribution of the treated vessel.
  3. Death within the first 30 days post index procedure (without other obvious cause) is considered a surrogate for stent thrombosis when angiography is not available.
Time Frame: 1-2 years
Population: To be analyzed in this secondary analysis, a subject needed to have an endpoint event between 1-2 years or sufficient follow-up through 2-years. There were 448 subjects that did not meet the criteria for this analysis.
Measure: Number; unit: percentage of participants
Arm/Group | TAXUS Libertē: Overall Enrolled Population
Number analyzed (Participants) | 3751
percentage of participants | 1.3

3. Secondary Outcome: Target Vessel Failure (TVF) for the Medically-Treated Diabetic Population
Description: Target vessel failure (TVF) for TAXUS Libertē Post-Approval Study medically-treated diabetic population. For pooled data from the TAXUS Liberté population, please see the citations
Time Frame: 12 months
Population: To be included, subject was a medically treated diabetic at the time of enrollment. Also, subjects met the following criteria: either a minimum number of days of follow-up of 335 days or an endpoint event up to 365 days post-stent implant procedure. There were 2945 subjects that did not meet the criteria for this analysis.
Measure: Number; unit: percentage of participants
Groups:
- Medically Treated Diabetic Population: Patients enrolled in the TAXUS Libertē Post-Approval Study with medically treated diabetes.
Arm/Group | Medically Treated Diabetic Population
Number analyzed (Participants) | 1254
percentage of participants | 6.1

4. Secondary Outcome: Rate of Major Adverse Cardiac and Cerebrovascular Events (MACCE)
Description: * MACCE defined as the composite of cardiac death, myocardial infarction, target vessel revascularization and stroke.
  * Binary rate
Time Frame: 6 months
Population: There were 67 patients that were not eligible for the 6-month analyses, as they did not meet the following criteria: either a minimum number of days of follow-up of 335 days or an endpoint event up to 365 days post-stent implant procedure.
Measure: Number; unit: percentage of participants
Groups:
- TAXUS Liberté: Overall Enrolled Population: Overall enrolled population of patients: received at least one TAXUS Liberté Paclitaxel-Eluting Coronary Stent System in routine clinical practice, in conjunction with the use of prasugrel and aspirin.
Arm/Group | TAXUS Liberté: Overall Enrolled Population
Number analyzed (Participants) | 4132
percentage of participants | 4.7

5. Secondary Outcome: Rate of Major Adverse Cardiac and Cerebrovascular Events (MACCE)
Description: as for outcome 4
Time Frame: 12 months
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | TAXUS Liberté: Overall Enrolled Population
Number analyzed (Participants) | 4059
percentage of participants | 7.8

6. Secondary Outcome: Rate of Major Adverse Cardiac & Cerebrovascular Events (MACCE): Study Stent Related
Description: MACCE defined as the composite of cardiac death, myocardial infarction, target vessel revascularization and stroke.
Time Frame: 6 months
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | TAXUS Liberté: Overall Enrolled Population
Number analyzed (Participants) | 4132
percentage of participants | 3.1

7. Secondary Outcome: Rate of Major Adverse Cardiac and Cerebrovascular Events (MACCE): Study Stent Related
Description: as for outcome 4
Time Frame: 12 months
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | TAXUS Liberté: Overall Enrolled Population
Number analyzed (Participants) | 4059
percentage of participants | 4.9

8. Secondary Outcome: Rate of Major Adverse Cardiac Events (MACE)
Description: * MACE defined as the composite of cardiac death, myocardial infarction and target vessel revascularization.
  * Binary rate
Time Frame: 6 months
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | TAXUS Liberté: Overall Enrolled Population
Number analyzed (Participants) | 4132
percentage of participants | 4.3

9. Secondary Outcome: Rate of Major Adverse Cardiac Events (MACE)
Description: as for outcome 8
Time Frame: 12 months
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | TAXUS Liberté: Overall Enrolled Population
Number analyzed (Participants) | 4059
percentage of participants | 7.3

10. Secondary Outcome: Rate of Major Adverse Cardiac Events (MACE): Study Stent Related
Description: as for outcome 8
Time Frame: 6 months
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | TAXUS Liberté: Overall Enrolled Population
Number analyzed (Participants) | 4132
percentage of participants | 3.1

11. Secondary Outcome: Rate of Major Adverse Cardiac Events (MACE): Study Stent Related
Description: as for outcome 8
Time Frame: 12 months
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | TAXUS Liberté: Overall Enrolled Population
Number analyzed (Participants) | 4059
percentage of participants | 4.9

12. Secondary Outcome: Rate of Target Vessel Failure (TVF)
Description: * Target vessel failure is defined as any revascularization of the target vessel, MI (Q- and non-Q wave) related to the target vessel, or death related to the target vessel.
  * Binary Rate
Time Frame: 6 months
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | TAXUS Liberté: Overall Enrolled Population
Number analyzed (Participants) | 4132
percentage of participants | 3.9

13. Secondary Outcome: Rate of Target Vessel Failure (TVF)
Description: as for outcome 12
Time Frame: 12 months
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | TAXUS Liberté: Overall Enrolled Population
Number analyzed (Participants) | 4059
percentage of participants | 6.4

14. Secondary Outcome: Rate of Cardiac Death or Myocardial Infarction (MI)
Description: - Binary Rate
Time Frame: 6 months
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | TAXUS Liberté: Overall Enrolled Population
Number analyzed (Participants) | 4132
percentage of participants | 1.4

15. Secondary Outcome: Rate of Cardiac Death or Myocardial Infarction (MI)
Description: - Binary Rate
Time Frame: 12 months
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | TAXUS Liberté: Overall Enrolled Population
Number analyzed (Participants) | 4059
percentage of participants | 2.1

16. Secondary Outcome: Rate of All Cause Death
Description: -Binary rate
Time Frame: 6 months
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | TAXUS Liberté: Overall Enrolled Population
Number analyzed (Participants) | 4132
percentage of participants | 0.7

17. Secondary Outcome: Rate of All Cause Death
Description: -Binary rate
Time Frame: 12 months
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | TAXUS Liberté: Overall Enrolled Population
Number analyzed (Participants) | 4059
percentage of participants | 1.4

18. Secondary Outcome: Rate of Cardiac Death
Description: -Binary rate
Time Frame: 6 months
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | TAXUS Liberté: Overall Enrolled Population
Number analyzed (Participants) | 4132
percentage of participants | 0.4

19. Secondary Outcome: Rate of Cardiac Death
Description: -Binary rate
Time Frame: 12 months
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | TAXUS Liberté: Overall Enrolled Population
Number analyzed (Participants) | 4059
percentage of participants | 0.9

20. Secondary Outcome: Rate of Cardiac Death: Study Stent Related
Description: -Binary rate
Time Frame: 6 months
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | TAXUS Liberté: Overall Enrolled Population
Number analyzed (Participants) | 4132
percentage of participants | 0.1

21. Secondary Outcome: Rate of Cardiac Death: Study Stent Related
Description: -Binary rate
Time Frame: 12 months
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | TAXUS Liberté: Overall Enrolled Population
Number analyzed (Participants) | 4059
percentage of participants | 0.1

22. Secondary Outcome: Rate of Myocardial Infarction (MI)
Description: -Binary rate
Time Frame: 6 months
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | TAXUS Liberté: Overall Enrolled Population
Number analyzed (Participants) | 4132
percentage of participants | 1.0

23. Secondary Outcome: Rate of Myocardial Infarction (MI)
Description: -Binary rate
Time Frame: 12 months
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | TAXUS Liberté: Overall Enrolled Population
Number analyzed (Participants) | 4059
percentage of participants | 1.4

24. Secondary Outcome: Rate of Myocardial Infarction (MI): Study Stent Related
Description: -Binary rate
Time Frame: 6 months
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | TAXUS Liberté: Overall Enrolled Population
Number analyzed (Participants) | 4132
percentage of participants | 0.9

25. Secondary Outcome: Rate of Myocardial Infarction (MI): Study Stent Related
Description: -Binary rate
Time Frame: 12 months
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | TAXUS Liberté: Overall Enrolled Population
Number analyzed (Participants) | 4059
percentage of participants | 1.0

26. Secondary Outcome: Rate of Target Vessel Reintervention (TVR)
Description: -Binary rate
Time Frame: 6 months
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | TAXUS Liberté: Overall Enrolled Population
Number analyzed (Participants) | 4132
percentage of participants | 3.3

27. Secondary Outcome: Rate of Target Vessel Reintervention (TVR)
Description: -Binary rate
Time Frame: 12 months
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | TAXUS Liberté: Overall Enrolled Population
Number analyzed (Participants) | 4059
percentage of participants | 5.8

28. Secondary Outcome: Rate of Target Vessel Reintervention (TVR): Study Stent Related
Description: -Binary rate
Time Frame: 6 months
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | TAXUS Liberté: Overall Enrolled Population
Number analyzed (Participants) | 4132
percentage of participants | 2.5

29. Secondary Outcome: Rate of Target Vessel Reintervention (TVR): Study Stent Related
Description: -Binary rate
Time Frame: 12 months
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | TAXUS Liberté: Overall Enrolled Population
Number analyzed (Participants) | 4059
percentage of participants | 4.3

30. Secondary Outcome: Rate of Stroke
Description: -Binary Rate
Time Frame: 6 months
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | TAXUS Liberté: Overall Enrolled Population
Number analyzed (Participants) | 4132
percentage of participants | 0.4

31. Secondary Outcome: Rate of Stroke
Description: -Binary Rate
Time Frame: 12 months
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | TAXUS Liberté: Overall Enrolled Population
Number analyzed (Participants) | 4059
percentage of participants | 0.5

32. Secondary Outcome: Rate of Major Bleeding
Description: * Major Bleeding defined as the composite of severe or moderate bleeding complication (based upon GUSTO classification).
  * Binary rate
Time Frame: 6 months
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | TAXUS Liberté: Overall Enrolled Population
Number analyzed (Participants) | 4132
percentage of participants | 2.3

33. Secondary Outcome: Rate of Major Bleeding
Description: as for outcome 32
Time Frame: 12 months
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | TAXUS Liberté: Overall Enrolled Population
Number analyzed (Participants) | 4059
percentage of participants | 3.6

34. Secondary Outcome: Rate of Stent Thrombosis (ARC Definite + Probable)
Description: * ARC - Academic Research Consortium
  * Binary rate
Time Frame: 6 months
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | TAXUS Liberté: Overall Enrolled Population
Number analyzed (Participants) | 4132
percentage of participants | 0.6

35. Secondary Outcome: Rate of Stent Thrombosis (ARC Definite + Probable)
Description: * ARC - Academic Research Consortium
  * Binary Rate
Time Frame: 12 months
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | TAXUS Liberté: Overall Enrolled Population
Number analyzed (Participants) | 4059
percentage of participants | 0.8

36. Secondary Outcome: Rate of Stent Thrombosis (Protocol Definition)
Description: -Binary rate
  The occurrence of any of the following:
  1. Clinical presentation of acute coronary syndrome with angiographic evidence of stent thrombosis:
     Angiographic documentation of acute complete occlusion (TIMI flow 0 or 1) of a previously successfully treated artery (TIMI flow 2 to 3 immediately after stent placement and diameter stenosis less than or equal to 30%) and/or Angiographic documentation of a flow limiting thrombus within or adjacent to a previously successfully treated lesion
  2. Acute MI in the distribution of the treated vessel.
  3. Death within the first 30 days post index procedure (without other obvious cause) is considered a surrogate for stent thrombosis when angiography is not available.
Time Frame: 6 months
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | TAXUS Liberté: Overall Enrolled Population
Number analyzed (Participants) | 4132
percentage of participants | 0.6

37. Secondary Outcome: Rate of Stent Thrombosis (Protocol Definition)
Description: as for outcome 36
Time Frame: 12 months
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | TAXUS Liberté: Overall Enrolled Population
Number analyzed (Participants) | 4059
percentage of participants | 0.9

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | TAXUS Liberté: Overall Enrolled Population
Serious Adverse Events (participants affected / at risk) | 1232/4199
Other Adverse Events (participants affected / at risk) | 293/4199
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TAXUS Liberté: Overall Enrolled Population (N=4199)
Angina pectoris (Cardiac disorders) | 253 (278)
Angina unstable (Cardiac disorders) | 100 (113)
Coronary artery disease (Cardiac disorders) | 77 (79)
Cardiac failure congestive (Cardiac disorders) | 48 (62)
Coronary artery stenosis (Cardiac disorders) | 50 (51)
Acute myocardial infarction (Cardiac disorders) | 46 (50)
Myocardial infarction (Cardiac disorders) | 45 (48)
Atrial fibrillation (Cardiac disorders) | 22 (26)
Coronary artery thrombosis (Cardiac disorders) | 21 (24)
Ventricular tachycardia (Cardiac disorders) | 16 (16)
Cardiac arrest (Cardiac disorders) | 15 (15)
Coronary artery dissection (Cardiac disorders) | 14 (15)
Ischaemic cardiomyopathy (Cardiac disorders) | 12 (12)
Myocardial ischaemia (Cardiac disorders) | 12 (12)
Bradycardia (Cardiac disorders) | 11 (11)
Ventricular fibrillation (Cardiac disorders) | 10 (10)
Acute coronary syndrome (Cardiac disorders) | 6 (6)
Cardiac failure (Cardiac disorders) | 6 (6)
Coronary artery occlusion (Cardiac disorders) | 5 (5)
Supraventricular tachycardia (Cardiac disorders) | 5 (5)
Atrioventricular block complete (Cardiac disorders) | 4 (4)
Sick sinus syndrome (Cardiac disorders) | 4 (4)
Arteriosclerosis coronary artery (Cardiac disorders) | 3 (3)
Cardiac failure chronic (Cardiac disorders) | 3 (3)
Cardiorespiratory arrest (Cardiac disorders) | 3 (3)
Cardiomyopathy (Cardiac disorders) | 3 (3)
Congestive myopathy (Cardiac disorders) | 3 (3)
Left ventricular dysfunction (Cardiac disorders) | 3 (3)
Arteriospasm coronary (Cardiac disorders) | 2 (2)
Atrioventricular block (Cardiac disorders) | 2 (2)
Cardiac tamponade (Cardiac disorders) | 2 (2)
Cardiogenic Shock (Cardiac disorders) | 2 (2)
Coronary artery perforation (Cardiac disorders) | 2 (2)
Mitral valve incompetence (Cardiac disorders) | 2 (2)
Palpitations (Cardiac disorders) | 2 (2)
Aortic Valve Stenosis (Cardiac disorders) | 1 (1)
Atrial tachycardia (Cardiac disorders) | 1 (1)
Atrioventricular block first degree (Cardiac disorders) | 1 (1)
Cardiac aneurysm (Cardiac disorders) | 1 (1)
Cardiac disorder (Cardiac disorders) | 1 (1)
Cardiac failure acute (Cardiac disorders) | 1 (1)
Cardiopulmonary failure (Cardiac disorders) | 1 (1)
Conduction Disorder (Cardiac disorders) | 1 (1)
Hypertensive heart disease (Cardiac disorders) | 1 (1)
Hypertrophic cardiomyopathy (Cardiac disorders) | 1 (1)
Intracardiac thrombus (Cardiac disorders) | 1 (1)
Left ventricular failure (Cardiac disorders) | 1 (1)
Microvascular angina (Cardiac disorders) | 1 (1)
Pericarditis (Cardiac disorders) | 1 (1)
Postural orthostatic tachycardia syndrome (Cardiac disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Stress cardiomyopathy (Cardiac disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
Ventricle Rupture (Cardiac disorders) | 1 (1)
Ventricular dysfunction (Cardiac disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 160 (183)
Chest pain (General disorders) | 20 (23)
Catheter site haemorrhage (General disorders) | 6 (7)
Adverse drug reaction (General disorders) | 6 (6)
Catheter site haematoma (General disorders) | 6 (6)
Death (General disorders) | 4 (4)
Asthenia (General disorders) | 3 (3)
Chest discomfort (General disorders) | 2 (2)
Impaired healing (General disorders) | 2 (2)
Multi-organ failure (General disorders) | 2 (2)
Pyrexia (General disorders) | 2 (2)
Catheter site discharge (General disorders) | 1 (1)
Catheter site pain (General disorders) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 51 (57)
Rectal haemorrhage (Gastrointestinal disorders) | 10 (10)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 9 (9)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 8 (8)
Gastritis (Gastrointestinal disorders) | 7 (7)
Pancreatitis (Gastrointestinal disorders) | 6 (6)
Pancreatitis acute (Gastrointestinal disorders) | 3 (5)
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 5 (5)
Small intestinal obstruction (Gastrointestinal disorders) | 5 (5)
Abdominal pain (Gastrointestinal disorders) | 4 (4)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 4 (4)
Haematemesis (Gastrointestinal disorders) | 4 (4)
Gastritis Haemorrhagic (Cardiac disorders) | 3 (3)
Peptic ulcer (Gastrointestinal disorders) | 3 (3)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2)
Colitis ischaemic (Gastrointestinal disorders) | 2 (2)
Diabetic gastroparesis (Gastrointestinal disorders) | 1 (2)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 2 (2)
Gastric ulcer (Gastrointestinal disorders) | 2 (2)
Gastritis erosive (Gastrointestinal disorders) | 2 (2)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 2 (2)
Impaired gastric emptying (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (2)
Retroperitoneal haematoma (Gastrointestinal disorders) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Abdominal hernia (Gastrointestinal disorders) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Colitis ulcerative (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Diverticulum (Gastrointestinal disorders) | 1 (1)
Diverticulum intestinal (Gastrointestinal disorders) | 1 (1)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1)
Entercolitis haemorrhagic (Gastrointestinal disorders) | 1 (1)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 (1)
Gastrointestinal ulcer (Gastrointestinal disorders) | 1 (1)
Gastrointestinal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1)
Hiatus hernia (Gastrointestinal disorders) | 1 (1)
Ileus paralytic (Gastrointestinal disorders) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 1 (1)
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 1 (1)
Lip haemorrhage (Gastrointestinal disorders) | 1 (1)
Localised intraabdominal fluid collection (Gastrointestinal disorders) | 1 (1)
Mallory-Weiss syndrome (Gastrointestinal disorders) | 1 (1)
Melaena (Gastrointestinal disorders) | 1 (1)
Obstruction gastric (Gastrointestinal disorders) | 1 (1)
Oesophageal rupture (Gastrointestinal disorders) | 1 (1)
Oesophageal ulcer (Gastrointestinal disorders) | 1 (1)
Oesophageal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1)
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 1 (1)
Pancreatic cyst (Gastrointestinal disorders) | 1 (1)
Pancreatic pseudocyst (Gastrointestinal disorders) | 1 (1)
Pacreatitis chronic (Gastrointestinal disorders) | 1 (1)
Peptic ulcer haemorrhage (Gastrointestinal disorders) | 1 (1)
Peptic ulcer perforation (Gastrointestinal disorders) | 1 (1)
Peritoneal haemorrhage (Gastrointestinal disorders) | 1 (1)
Peritonitis (Gastrointestinal disorders) | 1 (1)
Proctitis (Gastrointestinal disorders) | 1 (1)
Rectal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1)
Small intestine perforation (Gastrointestinal disorders) | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Pneumonia (Infections and infestations) | 29 (30)
Cellulitis (Infections and infestations) | 13 (15)
Bronchitis (Infections and infestations) | 7 (7)
Sepsis (Infections and infestations) | 7 (7)
Appendicitis (Infections and infestations) | 5 (5)
Diverticulitis (Infections and infestations) | 3 (5)
Abscess Limb (Infections and infestations) | 4 (4)
Gastroenteritis (Infections and infestations) | 3 (3)
Urinary Tract Infection (Infections and infestations) | 3 (3)
Cellulitis staphylococcal (Infections and infestations) | 1 (2)
Diabetic foot infection (Infections and infestations) | 2 (2)
Gangrene (Infections and infestations) | 2 (2)
Influenza (Infections and infestations) | 2 (2)
Lobar pneumonia (Infections and infestations) | 2 (2)
Osteomyelitis (Infections and infestations) | 2 (2)
Pneumonia staphylococcal (Infections and infestations) | 2 (2)
Septic shock (Infections and infestations) | 2 (2)
Sinusitis (Infections and infestations) | 2 (2)
Staphylococcal infection (Infections and infestations) | 2 (2)
Urosepsis (Infections and infestations) | 2 (2)
Wound infection (Infections and infestations) | 2 (2)
Abdominal wall access (Infections and infestations) | 1 (1)
Abdominal wall infection (Infections and infestations) | 1 (1)
Abscess intestinal (Infections and infestations) | 1 (1)
Bronchopneumonia (Infections and infestations) | 1 (1)
Bronchopulmonary aspergillosis allergic (Infections and infestations) | 1 (1)
Device related infection (Infections and infestations) | 1 (1)
Empyema (Infections and infestations) | 1 (1)
Fungal infection (Infections and infestations) | 1 (1)
Groin infection (Infections and infestations) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1)
Infected lymphocyle (Infections and infestations) | 1 (1)
Infected skin ulcer (Infections and infestations) | 1 (1)
Infection (Infections and infestations) | 1 (1)
Pneumonia bacterial (Infections and infestations) | 1 (1)
Pneumonia pneumococcal (Infections and infestations) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1)
Rectal abcess (Infections and infestations) | 1 (1)
Scrotal abcess (Infections and infestations) | 1 (1)
Sepsis syndrome (Infections and infestations) | 1 (1)
Staphylococcal bacteraemia (Infections and infestations) | 1 (1)
Steptococcal sepsis (Infections and infestations) | 1 (1)
Thrombophlebitis septic (Infections and infestations) | 1 (1)
Tracheobronchitis (Infections and infestations) | 1 (1)
Upper respiritory tract infection (Infections and infestations) | 1 (1)
Syncope (Nervous system disorders) | 20 (23)
Carotic artery stenosis (Nervous system disorders) | 13 (14)
Ischaemic stroke (Nervous system disorders) | 11 (11)
Transient ischaemic attack (Nervous system disorders) | 8 (8)
Presyncope (Nervous system disorders) | 6 (6)
Haemorrhage intracranial (Nervous system disorders) | 4 (4)
Dizziness (Nervous system disorders) | 3 (3)
Embolic stroke (Nervous system disorders) | 3 (3)
Subarachnoid haemorrhage (Nervous system disorders) | 3 (3)
Carotid sinus syndrome (Nervous system disorders) | 1 (2)
Cerebral haemorrhage (Nervous system disorders) | 2 (2)
Cerebral infarction (Nervous system disorders) | 2 (2)
Convulsion (Nervous system disorders) | 2 (2)
Neuropathy peripheral (Nervous system disorders) | 2 (2)
Paraesthesia (Nervous system disorders) | 2 (2)
Amnesia (Nervous system disorders) | 1 (1)
Anoxic encephalopathy (Nervous system disorders) | 1 (1)
Basilar artery thrombosis (Nervous system disorders) | 1 (1)
Brain stem infarction (Nervous system disorders) | 1 (1)
Burning sensation (Nervous system disorders) | 1 (1)
Carotic artery occlusion (Nervous system disorders) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1)
Cervicobrachial syndrome (Nervous system disorders) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1)
Facial palsy (Nervous system disorders) | 1 (1)
Guillain-Barre syndrome (Nervous system disorders) | 1 (1)
Hemianopia homonymous (Nervous system disorders) | 1 (1)
Hemiparesis (Nervous system disorders) | 1 (1)
Hepatic encephalopathy (Nervous system disorders) | 1 (1)
Hydrocephalus (Nervous system disorders) | 1 (1)
Hypertensive encephalopathy (Nervous system disorders) | 1 (1)
Lacunar infarction (Nervous system disorders) | 1 (1)
Lumbar radiculopathy (Nervous system disorders) | 1 (1)
Rapiculopathy (Nervous system disorders) | 1 (1)
Tarsal tunnel syndrome (Nervous system disorders) | 1 (1)
Thrombotic stroke (Nervous system disorders) | 1 (1)
Transient global amnesia (Nervous system disorders) | 1 (1)
Vertobasilar insufficiency (Nervous system disorders) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 8 (11)
Peripheral vascular disorder (Vascular disorders) | 10 (10)
Deep vein thrombosis (Vascular disorders) | 7 (8)
Hypertension (Vascular disorders) | 8 (8)
Hypotension (Vascular disorders) | 8 (8)
Intermittent claudication (Vascular disorders) | 6 (7)
Aortic stenosis (Vascular disorders) | 5 (5)
Orthostatic hypotension (Vascular disorders) | 5 (5)
Femoral arterial stenosis (Vascular disorders) | 4 (4)
Iliac artery stenosis (Vascular disorders) | 4 (4)
Peripheral ischaemia (Vascular disorders) | 4 (4)
Femoral artery occlusion (Vascular disorders) | 3 (3)
Haematoma (Vascular disorders) | 2 (2)
Hypertensive crisis (Vascular disorders) | 2 (2)
Malignant hypertension (Vascular disorders) | 2 (2)
Peripheral artery aneurysm (Vascular disorders) | 2 (2)
Vasospasm (Vascular disorders) | 1 (2)
Aortic aneurysm (Vascular disorders) | 1 (1)
Arterial fibrosis (Vascular disorders) | 1 (1)
Arterial haemorrhage (Vascular disorders) | 1 (1)
Arterial stenosis (Vascular disorders) | 1 (1)
Arterial stenosis limb (Vascular disorders) | 1 (1)
Arterial thrombosis limb (Vascular disorders) | 1 (1)
Arteriosclerosis (Vascular disorders) | 1 (1)
Blue toe syndrome (Vascular disorders) | 1 (1)
Haemorrhage (Vascular disorders) | 1 (1)
Hypertensive emergency (Vascular disorders) | 1 (1)
Iliac artery occlusion (Vascular disorders) | 1 (1)
Peripheral artery dissection (Vascular disorders) | 1 (1)
Subclavian artery stenosis (Vascular disorders) | 1 (1)
Venous stenosis (Vascular disorders) | 1 (1)
Chronic obstruction pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 13 (17)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 12 (15)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 10 (10)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 9 (9)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6 (7)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Status asthmaticus (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 16 (16)
Ankle fracture (Injury, poisoning and procedural complications) | 3 (4)
Contusion (Injury, poisoning and procedural complications) | 4 (4)
Hip fracture (Injury, poisoning and procedural complications) | 4 (4)
Subdural haematoma (Injury, poisoning and procedural complications) | 3 (4)
Overdose (Injury, poisoning and procedural complications) | 3 (3)
Post procedural myocardial infarction (Injury, poisoning and procedural complications) | 3 (3)
Anaemia postoperative (Injury, poisoning and procedural complications) | 2 (2)
Device malfunction (Injury, poisoning and procedural complications) | 2 (2)
Foot fracture (Injury, poisoning and procedural complications) | 2 (2)
Head injury (Injury, poisoning and procedural complications) | 2 (2)
Lower limb fracture (Injury, poisoning and procedural complications) | 2 (2)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 2 (2)
Rib fracture (Injury, poisoning and procedural complications) | 2 (2)
Anastamotic ulcer haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Burns third degree (Injury, poisoning and procedural complications) | 1 (1)
Contrast media reaction (Injury, poisoning and procedural complications) | 1 (1)
Device lead damage (Injury, poisoning and procedural complications) | 1 (1)
Facial bones fracture (Injury, poisoning and procedural complications) | 1 (1)
Fibula fracture (Injury, poisoning and procedural complications) | 1 (1)
Incision site haematoma (Injury, poisoning and procedural complications) | 1 (1)
Incision site pain (Injury, poisoning and procedural complications) | 1 (1)
Incisional hernia (Injury, poisoning and procedural complications) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 1 (1)
Mouth injury (Injury, poisoning and procedural complications) | 1 (1)
Poisoning (Injury, poisoning and procedural complications) | 1 (1)
Post procedural complication (Injury, poisoning and procedural complications) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1)
Scrotal haematoma (Injury, poisoning and procedural complications) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1)
Splenic rupture (Injury, poisoning and procedural complications) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1)
Traumatic lung injury (Injury, poisoning and procedural complications) | 1 (1)
Vascular procedure complication (Injury, poisoning and procedural complications) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 27 (28)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 5 (5)
Microcytic anaemia (Blood and lymphatic system disorders) | 2 (3)
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 2 (3)
Thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 (2)
Anaemic haemolytic autoimmune (Blood and lymphatic system disorders) | 1 (1)
Heparin-induced thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1)
Platelet aggregation inhibition (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 17 (18)
Renal failure (Renal and urinary disorders) | 7 (7)
Haematuria (Renal and urinary disorders) | 6 (6)
Nephrolithiasis (Renal and urinary disorders) | 3 (3)
Renal artery stenosis (Renal and urinary disorders) | 3 (3)
Nephrotic syndrome (Renal and urinary disorders) | 1 (2)
Pelvi-ureteric obstruction (Renal and urinary disorders) | 2 (2)
Renal failure chronic (Renal and urinary disorders) | 2 (2)
Renal impairment (Renal and urinary disorders) | 2 (2)
Calculus ureteric (Renal and urinary disorders) | 1 (1)
Cystitis haemorrhagic (Renal and urinary disorders) | 1 (1)
Urethral haemorrhagic (Renal and urinary disorders) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 7 (7)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 4 (5)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 4 (4)
Back Pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Costochondritis (Musculoskeletal and connective tissue disorders) | 2 (2)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 2 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Arthrofibrosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 (1)
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (5)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Benign neoplasm of bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Gastrointestinal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Hepatic cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Intestinal adenocarcenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lung adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lung adenocarcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lung squamous cell carcinoma stage 1 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lung squamous cell carcinoma stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lung squamous cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Pharyngeal cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Rectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Renal cancer carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 3 (3)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 2 (2)
Fluid overload (Metabolism and nutrition disorders) | 1 (2)
Gout (Metabolism and nutrition disorders) | 2 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 2 (2)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1)
Diabetic foot (Metabolism and nutrition disorders) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1)
Failure to thrive (Metabolism and nutrition disorders) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 1 (1)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1)
Obesity (Metabolism and nutrition disorders) | 1 (1)
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 7 (7)
Cholecystitis (Hepatobiliary disorders) | 5 (6)
Cholelithiasis (Hepatobiliary disorders) | 4 (4)
Biliary dyskinesia (Hepatobiliary disorders) | 2 (2)
Bile duct obstruction (Hepatobiliary disorders) | 1 (1)
Bile duct stenosis (Hepatobiliary disorders) | 1 (1)
Bile duct stone (Hepatobiliary disorders) | 1 (1)
Gallbladder disorder (Hepatobiliary disorders) | 1 (1)
Mental status changes (Psychiatric disorders) | 5 (5)
Alcohol withdrawal syndrome (Psychiatric disorders) | 2 (2)
Suicidal ideation (Psychiatric disorders) | 2 (2)
Anxiety (Psychiatric disorders) | 1 (1)
Completed suicide (Psychiatric disorders) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1)
Psychotic disorder (Psychiatric disorders) | 1 (1)
Cardiac enzymes increased (Investigations) | 4 (4)
Haemoglobin decreased (Investigations) | 4 (4)
Bacteria stool identified (Investigations) | 1 (1)
Blood glucose decreased (Investigations) | 1 (1)
Cardiac stress test abnormal (Investigations) | 1 (1)
Electrocardiogram abnormal (Investigations) | 1 (1)
Troponin increased (Investigations) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 4 (4)
Hypersensitivity (Immune system disorders) | 3 (3)
Menorrhagia (Reproductive system and breast disorders) | 3 (3)
Uterine prolapse (Reproductive system and breast disorders) | 1 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 (1)
Vaginal prolapse (Reproductive system and breast disorders) | 1 (1)
Haemorrhagic arteriovenous malformation (Congenital, familial and genetic disorders) | 2 (3)
Atrial septal defect (Congenital, familial and genetic disorders) | 2 (2)
Angioedema (Skin and subcutaneous tissue disorders) | 2 (2)
Skin ulcer (Skin and subcutaneous tissue disorders) | 2 (2)
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 2 (2)
Retinal artery occlusion (Eye disorders) | 1 (1)
Retinal detachment (Eye disorders) | 1 (1)
Primary hypothyroidism (Endocrine disorders) | 1 (1)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 12 (12)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TAXUS Liberté: Overall Enrolled Population (N=4199)
Myocardial infarction (Cardiac disorders) | 43 (43)
Coronary artery disease (Cardiac disorders) | 21 (21)
Coronary artery dissection (Cardiac disorders) | 7 (7)
Acute myocardial infarction (Cardiac disorders) | 2 (2)
Angina pectoris (Cardiac disorders) | 1 (1)
Angina unstable (Cardiac disorders) | 1 (1)
Coronary artery stenosis (Cardiac disorders) | 1 (1)
Coronary artery thrombosis (Cardiac disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 47 (47)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 9 (9)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 8 (8)
Gingival bleeding (Gastrointestinal disorders) | 4 (4)
Abdominal discomfort (Gastrointestinal disorders) | 3 (3)
Haematochezia (Gastrointestinal disorders) | 3 (3)
Melaena (Gastrointestinal disorders) | 3 (3)
Faeces discoloured (Gastrointestinal disorders) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 1 (1)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Adverse drug reaction (General disorders) | 20 (20)
Catheter site haematoma (General disorders) | 7 (7)
Catheter site haemorrhage (General disorders) | 2 (2)
Chest pain (General disorders) | 2 (2)
Catheter site discharge (General disorders) | 1 (1)
Catheter site related reaction (General disorders) | 1 (1)
Chest discomfort (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Puncture site haemorrhage (General disorders) | 1 (1)
Post-procedure myocardial infarction (Injury, poisoning and procedural complications) | 9 (9)
Contusion (Injury, poisoning and procedural complications) | 8 (8)
Animal scratch (Injury, poisoning and procedural complications) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1)
Tongue injury (Injury, poisoning and procedural complications) | 1 (1)
Vascular procedure complication (Injury, poisoning and procedural complications) | 1 (1)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1)
Venous injury (Injury, poisoning and procedural complications) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 19 (19)
Hypersensitivity (Immune system disorders) | 4 (4)
Haematoma (Vascular disorders) | 6 (6)
Haemorrhage (Vascular disorders) | 6 (6)
Arteriovenous fistula (Vascular disorders) | 1 (1)
Venous stenosis (Vascular disorders) | 1 (1)
Cardiac enzymes increased (Investigations) | 5 (5)
Troponin increased (Investigations) | 5 (5)
Bleeding time prolonged (Investigations) | 1 (1)
Blood creatine phosphokinase MB increased (Investigations) | 1 (1)
Haemoglobin decreased (Investigations) | 1 (1)
Haematuria (Renal and urinary disorders) | 10 (10)
Haemorrhage urinary tract (Renal and urinary disorders) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 3 (3)
Skin haemorrhage (Skin and subcutaneous tissue disorders) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 (1)
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 (1)
Rash generalise (Skin and subcutaneous tissue disorders) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 6 (6)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 2 (2)
Dizziness (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 1 (1)
Conjunctival haemorrhage (Eye disorders) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (2)
Hyphaema (Eye disorders) | 1 (1)
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 (1)
Haematospermia (Reproductive system and breast disorders) | 1 (1)
Menorrhagia (Reproductive system and breast disorders) | 1 (1)
Scrotal haematocoele (Reproductive system and breast disorders) | 1 (1)
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
During the term of the agreement and for a period of one year thereafter, the PI must submit to Boston Scientific each paper, summary, abstract or outline that he intends to present or publish relating to the study, and will not submit or present any proposed publication to a publisher or other party prior to the expiration of 45 days from the date such Proposed Publication is submitted to Boston Scientific.